CLINICAL TRIAL: NCT06096857
Title: A Phase 2b, Double-Blind, Randomized, Placebo-Controlled Trial of Cardamom and Topical Roseomonas in Atopic Dermatitis
Brief Title: Cardamom and Topical Roseomonas in Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10001677; 001677-I
Record Dates: First submitted 2023-10-21; First posted 2023-10-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-15

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Eczema; Atopic Dermatitis; Roseomonas; Cardamom; Itch; Rash
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus; Exanthema | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Roseomonas and Cardamom seeds
  Interventions: Drug: Roseomonas mucosa (RSM2015) and Cardamom seeds
- Placebo (Placebo Comparator): Sucrose
  Interventions: Drug: Placebo (sucrose)

INTERVENTIONS:
Drug: Roseomonas mucosa (RSM2015) and Cardamom seeds — Freeze dried packet to be reconstituted in water
  Arms: Active
Drug: Placebo (sucrose) — Freeze dried packet to be reconstituted in water
  Arms: Placebo

SUMMARY:
Background:

Atopic dermatitis (AD), also called eczema, is a chronic skin condition. AD can make skin dry and itchy, and sometimes it can lead to serious health problems, such as asthma, food allergies, eye infections, and sleep problems. No cure exists for AD. Researchers know that people with AD have different kinds of harmless bacteria on their skin than do people without AD. They want to see if adding a harmless bacteria (Roseomonas mucosa) to the skin can help people with AD.

Objective:

To test a skin treatment that contains R. mucosa and ground cardamom seeds in people with AD.

Eligibility:

People aged 2 years and older with AD.

Design:

All study visits will be remote. Participants will have 5 visits over about 7 months.

Participants will be screened. Researchers will review their AD and medical history.

Participants will receive a study product in the mail. The product comes as a powder in single-use packets. Participants will be shown how to mix the powder with water in a single-use spray vial. They will spray the solution onto their skin 2 to 3 times per week for 14 weeks.

Half of participants will receive the study powder. Half will receive a placebo; the placebo looks just like the study powder but contains no bacteria. They will not know which one they have.

During 3 study visits, participants will take a skin swab. They will receive supplies in the mail to rub a cotton swab on their skin and mail it back to the researchers.

Participants may opt to have pictures taken of their AD.

Participants will fill out 4 online questionnaires.

DETAILED DESCRIPTION:
Study Description:

This is a double-blind, randomized, phase 2b clinical trial for a topical formulation of a live biotherapeutic containing Roseomonas mucosa combined with ground cardamom seeds in a sucrose solution for patients with atopic dermatitis (AD). Participants will reconstitute the dried product in water and apply topically 2 or 3 times per week for 14 weeks. After 14 weeks, all interventions will cease, and participants will be followed for an additional 14 weeks to assess how long treatment effects last. During the course of study, we will assess disease severity (eg, itch, rash, and quality of life [QOL]) using a variety of AD assessments, ease of compliance with treatment, and changes in the microbiome profile of the skin. We hypothesize that topical treatment with Roseomonas mucosa, combined with ground cardamom seeds, will provide significantly more alleviation in AD symptoms than placebo, and that these effects will last beyond active treatment (due to the ability of the bacteria to colonize the patients' skin).

Primary Objective:

To determine if R mucosa combined with ground cardamom seeds can improve symptoms of AD in patients aged 2 and older, 14 weeks after treatment discontinuation.

Secondary Objective:

1. To determine if R mucosa combined with ground cardamom seeds can improve the Investigator s Global Assessment (IGA) in patients aged 2 and older, during active treatment as well as 7 weeks after treatment discontinuation, and at study completion.
2. To determine if R mucosa combined with ground cardamom seeds can improve the Numerical Rating Scale (NRS; both for average and worse severity over the 2-3 weeks prior to assessment) in patients aged 2 and older, during active treatment as well as 7 weeks after treatment discontinuation, and at study completion.
3. To determine if R mucosa combined with ground cardamom seeds can improve the SCORing Atopic Dermatitis (SCORAD) in patients aged 2 and older, during active treatment as well as 7 weeks after treatment discontinuation, and at study completion.
4. To determine if R mucosa combined with ground cardamom seeds can improve the Patient-Oriented Eczema Measure (POEM) in patients aged 2 and older, during active treatment as well as 7 weeks after treatment discontinuation, and at study completion.
5. To determine if effects of R mucosa combined with ground cardamom seeds on the symptoms of AD differ by levels of pollution near home of residence.
6. To determine if use of R mucosa permits less use of topical steroid treatments.
7. To determine the safety of R mucosa use.

Exploratory Objectives:

1. To determine if patients and caregivers using topical R mucosa understand the instructions and precautions for use.
2. To determine if topical R mucosa with cardamom seeds alters the skin microbiome profile during and after treatment.
3. To determine if topical R mucosa colonizes the skin of patients during use.

Primary Endpoint:

Proportion of participants achieving a 90% improvement in Eczema Area and Severity Index (EASI90; a measure of eczema rash) from baseline(week 0) to study completion (week 28).

Secondary Endpoints:

1. Proportion of adverse events (AEs).
2. Mean number of average weekly topical steroid use over the study follow up.
3. Change and percent change in IGA (a measure of eczema rash) from baseline (week 0) to: treatment completion (week 14), mid-follow-up (week 21), and study completion (week 28).
4. Change and percent change in EASI (a measure of eczema rash) from baseline (week 0) to: treatment completion (week 14), mid-follow-up (week 21), and study completion (week 28).
5. Change and percent change in NRS (subjective measure of itch) from baseline (week 0) to: treatment completion (week 14), mid-follow-up (week 21), and study completion (week 28).
6. Change and percent change in SCORAD (a combined metric of eczema itch, rash, QOL) from baseline (week 0) to: treatment completion (week 14), mid-follow-up (week 21), and study completion (week 28).
7. Change and percent change in QOL measures, POEM, from baseline (week 0) to: treatment completion (week 14), mid-follow-up (week 21), and study completion (week 28).
8. Association between improvement in EASI (a measure of eczema rash) from baseline (week 0) to study completion (week 28) and residence in high-pollution areas versus low-pollution areas.

Exploratory Endpoints:

1. Accuracy of identifying correct answers to questions about product applications and precautions.
2. Qualitative input regarding ease of use of product.
3. Presence of treatment strain of R mucosa as assessed by genetic detection (using polymerase chain reaction [PCR] primer).
4. Change in skin microbiome profile during and after treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all of the following criteria:

1. Aged >=2 years
2. Have a documented primary care provider near residence
3. Fluency in English (applicable to participant or caregiver who will be answering questionnaires)
4. Clinical diagnosis of AD, as defined by Hanifin and Rajka criteria, that has been present for >=3 months before the screening visit

   * Major Criteria: Must have >=3 basic features:

     * Pruritus
     * Typical morphology and distribution (flexural lichenification in adults, facial and extensor eruptions in infants and children)
     * Chronic or chronically relapsing dermatitis
     * Personal or family history of atopy (asthma, allergic rhinitis, AD)
   * Minor Criteria: Must have >=3 minor features:

     * Xerosis
     * Ichthyosis/palmar hyperlinearity, keratosis pilaris
     * Immediate (type 1) skin-test reactivity
     * Raised serum IgE
     * Early age of onset
     * Tendency toward cutaneous infections (especially Staphylococcus aureus and herpes simplex), impaired cell-mediated immunity
     * Tendency toward non-specific hand or foot dermatitis
     * Nipple eczema
     * Cheilitis
     * Recurrent conjunctivitis
     * Dennie-Morgan infraorbital fold
     * Keratoconus
     * Anterior subcapsular cataracts
     * Orbital darkening
     * Facial pallor, facial erythema
     * Pityriasis alba
     * Anterior neck folds
     * Itch when sweating
     * Intolerance to wool and lipid solvents
     * Perifollicular accentuation
     * Food intolerance
     * Course influenced by environmental or emotional factors
     * White dermographism, delayed blanch
5. EASI >5 and/or an IGA >=1 at time of enrollment.
6. Sexually active participants of childbearing potential must agree to use adequate methods of contraception from the screening visit continuously until 30 days after stopping treatment with the investigational product. Childbearing potential is defined for children as participants who have begun menstruating and for adults as participants who are not surgically sterile (hysterectomy and/or tubal ligation) or menopausal (age >=45 years plus no menses for 12 consecutive months without an alternative medical cause). Adequate contraception methods include: a barrier method (eg, condom use), oral contraceptive pill, hormonal patch or ring, hormonal injection, parenteral hormonal implant, or an intrauterine device.
7. Participants and parents/legal guardians (for minor participants) are willing and able to comply with all study visits and/or study-related procedures.
8. Participants/parents/guardians must have the ability to provide informed consent/assent as applicable.
9. Willingness to perform visits virtually.

EXCLUSION CRITERIA:

1. Previous treatment of AD:

   * Within 4 weeks prior to the baseline visit with any of the following:

     * Immunosuppressive or immunomodulating systemic drugs such as systemic corticosteroids, azathioprine, methotrexate, cyclosporine
     * Phototherapy or photochemotherapy for AD
   * Within 12 weeks prior to the baseline visit with any of the following having been newly initiated:

     * Topical steroids or topical calcineurin inhibitors
     * Janus kinase (JAK) inhibitors (oral or topical)
     * Dupilumab or any other biologic agent
     * Topical PDE4 inhibitor
     * Emollients containing ceramides, hyaluronic acid, urea or filaggrin degradation products.
     * Bleach baths
2. Active infection (chronic or acute) requiring treatment with systemic antibiotics, antivirals, or antifungals within 2 weeks before the baseline visit.
3. Superficial skin infection requiring topical treatment within 1 week of baseline visit.
4. Known or suspected history of immunosuppression or immunodeficiency.
5. Existence of indwelling central line.
6. Co-habitation with someone that has a known or suspected history of immunosuppression or immunodeficiency or has a central line.
7. Any clinically significant laboratory, history, or exam findings that, in the investigator's opinion, would suggest an increased risk to the participant.
8. Self-reported pregnancy or breastfeeding.
9. Menstruating females who have not menstruated within 6 weeks prior to screening. Participants who have an intrauterine device or implanted long-term contraceptive agent that prevents them from menstruating regularly will not be excluded.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
To determine if R mucosa combined with ground cardamom seeds can improve symptoms of AD in patients aged 2 and older, 14 weeks after treatment discontinuation. | From Baseline (week 0 to week 28)
  Proportion of participants achieving a 90% improvement in EASI90 (a measure of eczema rash) from baseline (week 0) to study completion (week 28).

SECONDARY OUTCOMES:
To determine if R mucosa combined with ground cardamom seeds can improve symptoms of AD in patients aged 2 and older, during active treatment as well as 7 weeks after treatment discontinuation. | Week 7 to week 28
  1. Proportion of AEs. 2. Proportion of participants using topical steroids over the course of the study.3. Change and percent change in IGA (a measure of eczema rash) from baseline (week 0) to: treatment completion (week 14), mid-washout (week 21) and study completion (week 28).4. Change and percent change in NRS (subjective measure of itch) from baseline (week 0) to: treatment completion (week 14), mid-washout (week 21), and study completion (week 28).5. Change and percent change in SCORAD (a combined metric of eczema itch, rash, QoL) from baseline (week 0) to: treatment completion (week 14), mid-washout (week 21), and study completion (week 28).6. Change and percent change in QOL measures, POEM, from baseline (week 0) to: treatment completion (week 14), mid-washout (week 21), and study completion (week 28).

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Myles, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All clinical data will be striped of PII and included in the publication. All microbiome data will be deposited in the appropriate databases.
Supporting Information: CSR
Time Frame: Upon publication.
Access Criteria: Public

REFERENCES:
- [Background] Li L, Han Z, Niu X, Zhang G, Jia Y, Zhang S, He C. Probiotic Supplementation for Prevention of Atopic Dermatitis in Infants and Children: A Systematic Review and Meta-analysis. Am J Clin Dermatol. 2019 Jun;20(3):367-377. doi: 10.1007/s40257-018-0404-3. PMID 30465329
- [Background] Mashiah J, Karady T, Fliss-Isakov N, Sprecher E, Slodownik D, Artzi O, Samuelov L, Ellenbogen E, Godneva A, Segal E, Maharshak N. Clinical efficacy of fecal microbial transplantation treatment in adults with moderate-to-severe atopic dermatitis. Immun Inflamm Dis. 2022 Mar;10(3):e570. doi: 10.1002/iid3.570. Epub 2021 Dec 20. PMID 34931478
- [Background] Myles IA, Castillo CR, Barbian KD, Kanakabandi K, Virtaneva K, Fitzmeyer E, Paneru M, Otaizo-Carrasquero F, Myers TG, Markowitz TE, Moore IN, Liu X, Ferrer M, Sakamachi Y, Garantziotis S, Swamydas M, Lionakis MS, Anderson ED, Earland NJ, Ganesan S, Sun AA, Bergerson JRE, Silverman RA, Petersen M, Martens CA, Datta SK. Therapeutic responses to Roseomonas mucosa in atopic dermatitis may involve lipid-mediated TNF-related epithelial repair. Sci Transl Med. 2020 Sep 9;12(560):eaaz8631. doi: 10.1126/scitranslmed.aaz8631. PMID 32908007
- [Background] Myles IA, Earland NJ, Anderson ED, Moore IN, Kieh MD, Williams KW, Saleem A, Fontecilla NM, Welch PA, Darnell DA, Barnhart LA, Sun AA, Uzel G, Datta SK. First-in-human topical microbiome transplantation with Roseomonas mucosa for atopic dermatitis. JCI Insight. 2018 May 3;3(9):e120608. doi: 10.1172/jci.insight.120608. PMID 29720571
- [Background] Nakatsuji T, Hata TR, Tong Y, Cheng JY, Shafiq F, Butcher AM, Salem SS, Brinton SL, Rudman Spergel AK, Johnson K, Jepson B, Calatroni A, David G, Ramirez-Gama M, Taylor P, Leung DYM, Gallo RL. Development of a human skin commensal microbe for bacteriotherapy of atopic dermatitis and use in a phase 1 randomized clinical trial. Nat Med. 2021 Apr;27(4):700-709. doi: 10.1038/s41591-021-01256-2. Epub 2021 Feb 22. PMID 33619370
- [Background] Yadav M, Chaudhary PP, D'Souza BN, Ratley G, Spathies J, Ganesan S, Zeldin J, Myles IA. Diisocyanates influence models of atopic dermatitis through direct activation of TRPA1. PLoS One. 2023 Mar 6;18(3):e0282569. doi: 10.1371/journal.pone.0282569. eCollection 2023. PMID 36877675
- [Background] Zeldin J, Chaudhary PP, Spathies J, Yadav M, D'Souza BN, Alishahedani ME, Gough P, Matriz J, Ghio AJ, Li Y, Sun AA, Eichenfield LF, Simpson EL, Myles IA. Exposure to isocyanates predicts atopic dermatitis prevalence and disrupts therapeutic pathways in commensal bacteria. Sci Adv. 2023 Jan 6;9(1):eade8898. doi: 10.1126/sciadv.ade8898. Epub 2023 Jan 6. PMID 36608129
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001677-I.html